CLINICAL TRIAL: NCT04407546
Title: Role of Children in the Transmission of SARS-CoV-2 in Households of Immunocompromised Persons
Brief Title: Role of Children in Transmission of COVID-19 to Immunocompromised Patients
Status: Terminated | Type: Observational
Why Stopped: enrollment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-000517; NCI-2020-03669 (Registry Identifier: CTRP)
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Immunosuppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects to provide biological specimens including nasal swabs, saliva and blood. Thereafter, participants will complete at-home nasal swab collections on a weekly basis for 6 months. If our research-use only SARS-CoV-2 test is positive, participants will be referred immediately to UCLA for medical attention and will be followed every 3 days with nasal swabs and saliva samples and weekly blood specimens and optional rectal swabs or fresh stool collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Families with Children: Families containing an immunocompromised individual that have children in the family setting.
- Famlies without children: Families containing an immunocompromised individual that do not have children in the family setting.

SUMMARY:
This is a study of immunosuppressed individuals living in households with and without children to assess the role of household contact with children in the transmission of SARSCoV-2 to immunocompromised individuals. Through careful collection of epidemiological data in combination with biological specimens, risk factors for SARS-CoV-2 in immunocompromised individuals will be identified. During the initial visits, informed consent will be obtained and consented participants will complete an initial questionnaire and provide biological specimens including nasal swabs, saliva and blood. Thereafter, participants will complete at-home saliva collections and questionnaires on a weekly basis for 6 months. If our research-use only SARS-CoV-2 test is positive, participants will be referred immediately for medical attention and will be followed every 3 days with nasal swabs and saliva samples and weekly blood specimens and optional rectal swabs or fresh stool collection. Additionally, participants will be contacted by telephone at 1 year for follow-up.

DETAILED DESCRIPTION:
This is a prospective, longitudinal cohort study of immunosuppressed patients living in households with and without children to assess the role of household contact with children in the transmission of SARS-CoV-2 to immunocompromised patients. This study will be enrolling both pediatric and adult patients who are immunosuppressed, as well as their household members who agree to participate. Through careful collection of epidemiological data in combination with biological specimens, risk factors for SARS- CoV-2 in immunocompromised patients will be identified. During the initial study visit, informed consent will be obtained, the study questionnaire will be completed and the participant will provide biological specimens including nasal mid-turbinate swabs, saliva and blood. Thereafter, participants will complete at-home saliva collections and questionnaires on a weekly basis for 6 months. If our research-use only SARS-CoV-2 test is positive, participants will be referred immediately to University of California at Los Angeles(UCLA) Health for medical attention and will be followed every 3 days with nasal swabs and saliva samples, and weekly blood specimens and optional rectal swabs or fresh stool collection. Biological specimen and questionnaire follow-up will occur for 6 months for uninfected participants or until the of end of viral shedding and immunologic profiling for patients infected with SARS-CoV-2, whichever is longer. All participants will be followed at 6 months with the same baseline measurements and then participants will be contacted by telephone at 1 year.

The clinical data and biological specimens collected in this initial study will provide will inform and allow future studies of clinical outcomes, viral characteristics, and immune responses to SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised patient followed at UCLA Health
* Immunocompromised patient >1 day old to <60 years of age
* Patient with a diagnosis of breast, lung, or colorectal cancers, lymphoma, acute/chronic leukemia, multiple myeloma, or other solid tumors and are receiving chemotherapy
* Patients who have received a hematopoietic stem cell transplantation within the last year
* Patients who have received a solid organ transplantation within the last year

Exclusion Criteria:

* Immunocompromised patients with positive SARS-CoV-2 test prior to study enrollment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Potentially eligible patients will be identified through examination of the electronic health record to identify patients receiving chemotherapy who are potentially eligible and could be approached for participation. Invitation to the study will occur through the MyChart portal or paper mailing letter, and those who are interested in participation will contact the research coordinator by phone or e-mail to undergo telephone screening for study eligibility. In addition, the research team member will explain the study objectives and procedures, and assess interest in participation. Pediatric recruitment of solid organ and hematopoietic stem cell transplantation patients will be done in collaboration with those respective primary pediatric subspecialist. The pediatric subspecialist teams will identify the patients who meet the inclusion criteria and will send the recruitment letter directly to the parents or patients if >18 years old via MyChart or paper mailed letter.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
To define the role of household contact with children or siblings in the transmission of SARS-CoV-2 to immunocompromised patients. | up to one year
  Measure the incidence of transmission of SARS-CoV-2 to immunocompromised patients in households with children compared to households without children

SECONDARY OUTCOMES:
To characterize secondary cases of SARS-CoV-2 in immunocompromised participants | up to one year
  Measure the rate of serology conversion of SARS-CoV-2 to immunocompromised patients in households with children compared to households without children
To describe the exposure factors such as pets and travel and how those factors are related to immunocompromised patients to estimate risk profiles by household characteristics | up to one year
  Measure the rates of exposures to the following risk factors: persons with positive SARS-CoV-2 PCR test, pets, previous travel to the incidence of transmission of SARS-CoV-2 to immunocompromised patients in households with children compared to households without children.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Aldrovandi, M.D., Principal Investigator — University of Califiornia at Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided